CLINICAL TRIAL: NCT00765193
Title: The Impact of Total Body Skin Examination on Skin Cancer Detection
Acronym: TBSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Prof. Rainer Hofmann-Wellenhof, Department of Dermatology; Medical University of Graz-Austria
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-175 ex 07/08
Record Dates: First submitted 2008-08-14; First posted 2008-10-02 (Estimated); Results first posted 2010-04-15 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Melanoma; Basal Cell Carcinoma; Squamous Cell Carcinoma; Merkel Cell Carcinoma; Skin Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Carcinoma, Merkel Cell; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Skin cancer screening (Other)
  Interventions: Other: Inspection of covered areas

INTERVENTIONS:
Other: Inspection of covered areas — Clinicans performed a two-step examination for skin cancer, with clinical examination of individual lesions was aided by the use of dermoscopy, as needed. In the first step, physicians performed inspection of problem areas and uncovered areas only, and lesions suggestive of melanoma or non-melanoma skin cancer were noted. In the second step, TBSE was performed. Following both examinations, lesions suggestive of melanoma or non-melanoma skin cancer were excised or biopsied. Histopathologic diagnosis was recorded for each of the biopsied or excised lesions.
  Other Names: Inspection of problem areas

SUMMARY:
This will be a study where all patients will undergo a two-step procedure:

Step 1 - Physicians examine the problem area of skin ONLY and record result. Step 2 - Physicians perform TBSE and record result. Eventual lesions suggestive of melanoma and non-melanoma skin cancers will be recorded after step 1 or step 2 examination and will be finally biopsied and histopathologically diagnosed. Exceptions to biopsy may include patients with multiple non-melanoma skin cancers (e.g. actinic keratoses or basal cell carcinomas).

Each center will be provided with an electronic data sheet for patients record, or alternatively, with a paper record form.

Endpoints of the study are new parameters concerning the standard of care for skin cancer screening. We expect to conclude that TBSE enables clinicians discovering an increased number of skin cancers thus resulting in earlier detection.

DETAILED DESCRIPTION:
Clinicans performed a two-step examination for skin cancer, with clinical examination of individual lesions was aided by the use of dermoscopy, as needed. In the first step, physicians performed inspection of problem areas and uncovered areas only, and lesions suggestive of melanoma or non-melanoma skin cancer were noted. In the second step, TBSE was performed. Following both examinations, lesions suggestive of melanoma or non-melanoma skin cancer were excised or biopsied. Histopathologic diagnosis was recorded for each of the biopsied or excised lesions.

Statistical analysis: We calculated absolute risks as the proportion of individuals with the target disease divided by all individuals at risk. The number needed to examine was calculated by dividing the individuals at risk by the numbers of individuals with the target disease. Confidence intervals for proportions were calculated using standard formulas based on the binomial distribution. Chi square tests were used for comparison of proportions.

Continuous variables are presented as mean and standard deviation (SD) unless otherwise specified. For univariate and multivariate analyses we used odds ratios derived from logistic regression to estimate relative risks and their confidence intervals. All p-values reported are 2-tailed. Statistical significance is defined as P <0.05. Statistical analysis was performed using SPSS software, version 16.0 (SPSS, Chicago, Ill, US).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive, unselected adult (18 years or more) patients with any skin disorders. Skin disorder must be localized on a limited body area and should NOT require total body skin examination (TBSE) to be diagnosed and/or treated.

Exclusion Criteria:

* Patients who ask for or need TBSE as the main reason for consultation. A patient must be also excluded if a significant part of the body should be undressed for diagnosis and/or treatment (i.e. if the shirt or trousers should be removed for diagnosis and/or treatment, then the patient must be excluded).
* patients under the age of 18 years.
* patients who do not agree to get TBSE.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14381 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Hofmann-Wellenhof, Prof., Principal Investigator — Medical University of Graz, Austria; Giuseppe Argenziano, Prof., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Medical University of Graz-Austria: Department of Dermatology, Graz, Austria

REFERENCES:
- [Derived] Argenziano G, Zalaudek I, Hofmann-Wellenhof R, Bakos RM, Bergman W, Blum A, Broganelli P, Cabo H, Caltagirone F, Catricala C, Coppini M, Dewes L, Francia MG, Garrone A, Turk BG, Ghigliotti G, Giacomel J, Gourhant JY, Hlavin G, Kukutsch N, Lipari D, Melchionda G, Ozdemir F, Pellacani G, Pellicano R, Puig S, Scalvenzi M, Sortino-Rachou AM, Virgili AR, Kittler H. Total body skin examination for skin cancer screening in patients with focused symptoms. J Am Acad Dermatol. 2012 Feb;66(2):212-9. doi: 10.1016/j.jaad.2010.12.039. Epub 2011 Jul 14. PMID 21757257

RESULTS

PARTICIPANT FLOW:
Groups:
- Skin Cancer Screening: Physicians examine, first, the problem area of skin and record result, and second, the full body and record result.
Period: Problem Area Examination
Arm/Group | Skin Cancer Screening
Started | 14381
Completed | 14381
Not Completed | 0
Period: Full Body Examination
Arm/Group | Skin Cancer Screening
Started | 14381
Completed | 14381
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Skin Cancer Screening
Number analyzed (Participants) | 14381
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11027
  >=65 years | 3354
Age Continuous [Mean (Standard Deviation); unit: years] | 49.4 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7984
  Male | 6397
Region of Enrollment [Number; unit: participants]
  Austria | 997
  Italy | 7381
  Brazil | 2010
  France | 999
  Argentina | 1001
  Netherlands | 787
  Spain | 179
  Turkey | 984
  Australia | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Suspicious Tumors Detected After Inspection of Problem Area and Inspection of the Full Body.
Time Frame: one year
Population: From a population of patients with various skin conditions, participants were considered for inclusion only if aged 18 years or more, and if suffering from focused skin complaints. Patients with diffuse skin complaints were excluded.
Measure: Number; unit: participants
Arm/Group | Problem Area Examination | Full Body Examination
Number analyzed (Participants) | 14381 | 14381
participants | 810 | 631
Statistical Analysis 1: Comparison: Problem Area Examination vs Full Body Examination; The primary outcomes were the calculation of the absolute and relative risks of missing a skin cancer when TBSE is not performed, as well as the number of patients needed to examine by TBSE to find a skin cancer. The secondary outcome was to assess the magnitude of false-positive results obtained by TBSE; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 2.36, 95% CI [2.12 to 2.62]

2. Secondary Outcome: Whether a Systematic Screening is Related to a Higher Number of Unnecessary Excisions of Benign Skin Tumors Detected During the Screening.
Time Frame: one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: No adverse events were collected for this study
Arm/Group | Skin Cancer Screening
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No